CLINICAL TRIAL: NCT02366130
Title: Phase II Trial of Ra-223 Dichloride in Combination With Hormonal Therapy and Denosumab in the Treatment of Patients With Hormone-Positive Bone-Dominant Metastatic Breast Cancer
Brief Title: Trial of Ra-223 Dichloride in Combination With Hormonal Therapy and Denosumab in the Treatment of Patients With Hormone-Positive Bone-Dominant Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0508; NCI-2015-00508 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Hormone-positive bone-dominant metastatic breast cancer; Ra-223 dichloride; Xofigo; Radium-223 chloride; Radium-223 dichloride; Alpharadin; Denosumab; AMG 162; Prolia; Hormone therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — radium Ra 223 dichloride; Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ra-223 dichloride + Denosumab (Experimental): Ra-223 dichloride 55 kBq/kg administered as a bolus intravenous (IV) injection (over 1 minute) through a secure in-dwelling catheter on day 1 of the study and then every four weeks thereafter for 6 cycles.
  Denosumab 120 mg by subcutaneous (SC) injections on Day 1 of Cycles 2-5.
  A single hormonal agent (ie, Tamoxifen or Aromatase Inhibitor or Fulvestrant) administered daily while on study. Physician to decide what type of hormone therapy participant will receive.
  Interventions: Drug: Ra-223 dichloride; Drug: Denosumab; Drug: Hormone Therapy

INTERVENTIONS:
Drug: Ra-223 dichloride — 55 kBq/kg by vein on Day 1 of each 28 day cycle, and then every four weeks thereafter for 6 cycles.
  Other Names: Xofigo; Radium-223 chloride; Radium-223 dichloride; Alpharadin
Drug: Denosumab — 120 mg by subcutaneous (SC) injections on Day 1 of Cycles 2-5.
  Other Names: AMG 162; Prolia
Drug: Hormone Therapy — A single hormonal agent administered daily while on study. Physician to decide what type of hormone therapy participant will receive.

SUMMARY:
The goal of this clinical research study is to learn if Xofigo® (also called Ra-223 dichloride) combined with hormone therapy and denosumab can help to control breast cancer that has spread to the bones and/or bone marrow. The safety of this study drug combination will also be studied.

This is an investigational study. Denosumab and the hormone therapies used in this study are FDA-approved and commercially available for the treatment of metastatic breast cancer. Ra-223 dichloride is FDA-approved and commercially available for the treatment of bone metastases. It is considered investigational to use the combination of Ra-223 dichloride, hormone therapy and denosumab to treat patients with bone cancer that has spread to the bones.

The study doctor can explain how the study drugs are designed to work.

Up to 36 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive Ra-223 dichloride by vein over no more than 1 minute on Day 1 of each 28-day study cycle.

You will also receive denosumab as an injection under the skin on Day 1 of Cycles 1- 6.

You will also receive hormone therapy while on study. Your doctor will discuss with you what type of hormone therapy you will have, how it will be given, and its risks.

Study Visits:

On Day 1 of Cycle 1, blood (about 2 teaspoons) will be drawn for routine tests.

On Day 1 of Cycles 2-5:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.

On Day 1 of Cycle 6:

* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* Blood (about 3 tablespoons) will be drawn for biomarker testing, including genetic biomarkers.
* Blood (about 5 teaspoons) will be drawn to test for CTCs, tumor markers, and genetic testing.
* You will have a PET-CT scan and a bone scan to check the status of the disease. If the doctor thinks it is needed, you will also have an MRI.

Length of Study Participation:

You may continue taking the study drugs for up to 6 cycles. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation will be over after the end-of-study visit.

End-of-Study Visit:

After your last dose of study drug:

* You will have a physical exam.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* Blood (about 3 tablespoons) will be drawn for biomarker testing, including genetic biomarkers.
* Blood (about 5 teaspoons) will be drawn to test for CTCs, tumor markers, and genetic testing.
* You will have a PET-CT scan and either a bone scan or a CT scan to check the status of the disease. If the doctor thinks it is needed, you will also have an MRI.
* If the doctor thinks it is needed, you will have a bone marrow aspiration/biopsy to check the status of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IV breast cancer with metastases to the bone and/or bone marrow.
2. Pathological or radiographically confirmation of metastases to the bone and/or bone marrow. (The definition of radiologic diagnosis of bone metastasis is based on typical and highly reliable imaging findings in studies such as bone scan (new or multiple TC99m positive lesions), PET/CT (new or multiple FRG positive lesions), and MRI (typical T1w replacement, T2w positive and T1 plus contrast media positive) for bone metastasis with 2 or more lesions. If the bone metastasis is highly suspected or not well defined by imaging, bone biopsy is necessary for confirmation.)
3. Visible uptake in at least one lesion on bone scanning prior to radium therapy.
4. No limit in number of prior hormonal agents in metastatic breast cancer; only one prior chemotherapy is allowed in metastatic setting. Anti-HER2 targeting therapy, CDK4/6 inhibitor, other targeted therapy (e.g., mTOR or PI3K inhibitor) in combination with hormonal treatment will be counted as one hormonal agent. Any anti-HER2 targeting therapy in combination with chemotherapy will not be counted as one additional treatment.
5. Breast tumors with hormone receptor positive disease (ER+/PR+, ER+/PR- regardless of HER2 status).
6. ECOG performance score of 0, 1.
7. Age =/> 18 years.
8. All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v4.0 Grade 1 or less at the time of signing the Informed Consent Form (ICF).
9. Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 6 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
10. Acceptable hematology and serum biochemistry screening values: White Blood Cell Count (WBC) =/> 3,000/mm3 Absolute Neutrophil Count (ANC) =/> 1,500/mm3 Platelet (PLT) count =/> 100,000/mm3 Hemoglobin (HGB) =/> 10 g/dl Total bilirubin level </=2.0 x institutional upper limit of normal (ULN) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </= 3.0 x ULN Creatinine </= 1.5 x ULN
11. Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.

Exclusion Criteria:

1. Following breast cancer disease conditions are not eligible: A) Single Bone Lesion. B)Two or more visceral metastasis C) Single visceral lesion < 2cm without any laboratory changes or clinical symptoms due to the metastatic lesion is permitted. D)Presence of brain metastases E) Imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). T F) Impending fracture, spinal cord compression, and/or potentially unstable compression fracture of vertebral body with possibility of cord compression. G) Life expectancy severely limited by concomitant illness (less than 12 months). H) Concurrent external beam radiation therapy to non target lesion is permitted.
2. Following prior treatments are not eligible. A) Use of any investigational agent within 30 days preceding enrollment. B) Treatment with cytotoxic chemotherapy within previous 4 weeks C) Failure to achieve </= Grade 2 AE resolution from cytotoxic chemotherapy administered more than 4 weeks previous (however, ongoing neuropathy is permitted). D) Received systemic therapy with radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188, or Ra-223 dichloride) for the treatment of bony metastases.
3. Following medical conditions are not eligible. A) Other malignancy treated within the last 3 years (except non melanoma skin cancer or low-grade superficial bladder cancer or cervical dysplasia) B) Any other serious illness or medical condition, such as but not limited to: Any infection =/> National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 Grade 2. C) Cardiac failure New York Heart Association (NYHA) III or IV. D) Crohn's disease or ulcerative colitis-Bone marrow dysplasia or Myelodysplastic syndrome.
4. Women who are pregnant or breast-feeding. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
5. Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
6. Major surgery within 30 days prior to start of study drug.
7. Excluded therapies and medications, previous and concomitant: A) Concurrent anti-cancer therapy (chemotherapy, surgery, immunotherapy, biologic therapy, anti-HER 2 targeting therapies, or tumor embolization) other than Ra 223 dichloride. Concurrent external beam radiation therapy is permitted.B) Prior use of Ra-223 dichloride. C) Concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 4 weeks of trial entry (signing of the informed consent form).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ueno NT, Tahara RK, Fujii T, Reuben JM, Gao H, Saigal B, Lucci A, Iwase T, Ibrahim NK, Damodaran S, Shen Y, Liu DD, Hortobagyi GN, Tripathy D, Lim B, Chasen BA. Phase II study of Radium-223 dichloride combined with hormonal therapy for hormone receptor-positive, bone-dominant metastatic breast cancer. Cancer Med. 2020 Feb;9(3):1025-1032. doi: 10.1002/cam4.2780. Epub 2019 Dec 18. PMID 31849202
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participating subjects must sign the consent document pertaining to the study and meet all the eligibility criteria as mentioned in the protocol, before initiating on the study treatment. This study was conducted at the University of Texas MD Anderson Cancer Center. All patients received at least one dose of Radium-223 and thus were evaluable for toxicity and disease control rate at 9 months.
Groups:
- Ra-223 Dichloride + Denosumab: Ra-223 dichloride 55 kBq/kg administered as a bolus intravenous (IV) injection (over 1 minute) through a secure in-dwelling catheter on day 1 of the study and then every four weeks thereafter for 6 cycles.
  Denosumab 120 mg by subcutaneous (SC) injections on Day 1 of Cycles 2-5.
  A single hormonal agent (ie, Tamoxifen or Aromatase Inhibitor or Fulvestrant) administered daily while on study. Physician to decide what type of hormone therapy participant will receive.
  Ra-223 dichloride: 55 kBq/kg by vein on Day 1 of each 28 day cycle, and then every four weeks thereafter for 6 cycles.
  Denosumab: 120 mg by subcutaneous (SC) injections on Day 1 of Cycles 2-5.
  Hormone Therapy: A single hormonal agent administered daily while on study. Physician to decide what type of hormone therapy participant will receive.
Period: Overall Study
Arm/Group | Ra-223 Dichloride + Denosumab
Started | 45
Completed | 36
Not Completed | 9
Not completed — Withdrawal by Subject | 3
Not completed — Ineligible | 6

BASELINE CHARACTERISTICS:
Arm/Group | Ra-223 Dichloride + Denosumab
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 58 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Control Rate at 9 Months
Description: Disease control rate is defined as the rate of the patients at that time with clinically complete or partial response or stable disease.
Time Frame: 9 months from receiving the first dose of Radium-223
Population: 1 patient was lost to FU between 6 and 9 months from first dose of Radium -223
Measure: Count of Participants; unit: Participants
Arm/Group | Ra-223 Dichloride + Denosumab
Number analyzed (Participants) | 35
Participants | 35

2. Primary Outcome: The Number of Participants With Disease Control Rate at 6 Months
Description: as for outcome 1
Time Frame: 6 months from receiving the first dose of Radium-223
Measure: Count of Participants; unit: Participants
Arm/Group | Ra-223 Dichloride + Denosumab
Number analyzed (Participants) | 36
Participants | 21

ADVERSE EVENTS:
Time Frame: adverse events were collected from First dose of Ra-223 up to 9 months
Arm/Group | Ra-223 Dichloride + Denosumab
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 28/36
Other Adverse Events (participants affected / at risk) | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ra-223 Dichloride + Denosumab (N=36)
Bone pain (Musculoskeletal and connective tissue disorders) | 28 (28)
Fatigue (General disorders) | 15 (15)
Nausea (Gastrointestinal disorders) | 13 (13)
AST/ALT elevation (Hepatobiliary disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Headache (Nervous system disorders) | 7 (7)
Hyperglycemia (Endocrine disorders) | 7 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (6)
Flu-like symptoms (General disorders) | 6 (6)
Hot Flashes (General disorders) | 5 (5)
Arthralgia (Infections and infestations) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4)
Lymphocytopenia (Blood and lymphatic system disorders) | 10 (10)
Neutropenia (Blood and lymphatic system disorders) | 9 (9)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT02366130/Prot_SAP_000.pdf